CLINICAL TRIAL: NCT02686203
Title: A Feasibility Study to Evaluate the Effectiveness of Low Level Laser Therapy Combined With Acupuncture as Palliative Treatment of Patients With Various Solid Malignancies Who Are no Longer Candidates for Active Oncological Therapies
Brief Title: Evaluate the Effectiveness of Low Level Laser Therapy (LLT) Combined With Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erika Carmel ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GD-IP-101
Record Dates: First submitted 2016-02-09; First posted 2016-02-19 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B-Cure Laser Pro and needles (Experimental): Treatment will consist of acupuncture applied by a combination of B-Cure Laser Pro, an approved handheld, portable device emitting low level laser, and needles using two to four acupoints (The Investigational Therapy).
  The Investigational Therapy will be administered by a treating therapist designated by the Sponsor who is experienced in employing the treatment.
  Interventions: Device: B-Cure Laser Pro and needles

INTERVENTIONS:
Device: B-Cure Laser Pro and needles — Treatment will consist of acupuncture applied by a combination of B-Cure Laser Pro, an approved handheld, portable device emitting low level laser, and needles using two to four acupoints (The Investigational Therapy).
  The Investigational Therapy will be administered by a treating therapist designated by the Sponsor who is experienced in employing the treatment

SUMMARY:
evaluating The Investigational Therapy effects on quality of life, pain and patient's clinical status in adult cancer patients with solid tumors who are no longer candidates for active oncological therapies.

DETAILED DESCRIPTION:
evaluating The Investigational Therapy effects on quality of life, pain and patient's clinical status in adult cancer patients with solid tumors who are no longer candidates for active oncological therapies.

Eligible patients will be enrolled into the study and receive at least two 20-min treatment sessions, 2 to 12 weeks apart, with the Investigational Therapy on healthy body tissue (i.e. non-tumor region) of back of the hand and/or foot. Number of treatment sessions and treatment frequency will be individualized per patient depending on patient's status as well as per the discretion of the treating therapist, who is specialized and experienced with using the Investigational Therapy. Patients will be assessed for quality of life, pain and patient's clinical status according to acceptable clinical evaluations.

If at any time after the start of this study, it will be decided to initiate active oncological treatment, the principal investigator or designee will inform the Sponsor. The Sponsor will decide if the patient will stay or be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 to 70 years of age diagnosed with cancer (with or without metastasis) including but not limited to breast, ovarian, cervical, uterine, renal, bladder, gastric, pancreas, lung, thyroid, colorectal, small and large intestine, testicle and prostate cancer who have either

   1. failed standard treatment for their type of cancer
   2. decline standard treatment and interested in non-invasive treatment or change in life style
   3. have time to decide on treatment options and interested in non-invasive treatment
2. Confirm cancer diagnosis using biopsy, biomarkers or imaging (PET/CT, MRI, CT, Ultrasound, etc.)
3. Karnofsky performance status score of at least 60% for lung cancer and at least 50% for all other cancers at the screening visit
4. Life expectancy of at least 12 weeks
5. Patients must have adequate organ function as defined below:

   1. AST (SGOT)/ALT(SGPT) <3x upper limit of normal (ULN).
   2. Serum creatinine <2.0 mg/dL.
   3. Serum bilirubin <3 mg/dL
6. Signed written informed consent to participate in the study independently by patient.
7. Ability to comply with the requirements of the study.

Exclusion Criteria:

1. Participation in an interventional investigational trial within 30 days of the screening visit.
2. Receipt of chemotherapy or radiotherapy within 1 month of the screening visits
3. Patients with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study or interfere with the evaluation of the investigational therapy effect (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive cardiac failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
4. Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator or the sponsor, of interfering with the conduct of the study.
5. who are likely to be non-compliant or uncooperative during the study. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life using World Health Organization Quality of Life questionnaire (WHOQoL-BREF) | 3 months
  After treatment Quality of life will be measured by using World Health Organization Quality of Life questionnaire (WHOQoL-BREF)
Quality of life using patient questionnaire Karnofsky performance status | 3 months
  After treatment Quality of life will be measured by using patient questionnaire Karnofsky performance status

SECONDARY OUTCOMES:
Self-reported pain perception using SF-MPQ | 3 months
  After treatment pain perception will be measured by using Self-reported pain perception using SF-MPQ
Self-reported pain perception using pain diagram | 3 months
  After treatment pain perception be measured by using pain diagram

OTHER OUTCOMES:
Safety Outcome - Adverse events related to Investigational therapy | 3 months
  Adverse events related to Investigational therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ido Wolf, MD, Principal Investigator — head of Medical Oncology Unit Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: No